CLINICAL TRIAL: NCT05136547
Title: Comparative Study of the Efficacy of Biologics vs Usual Treatment on OCS Reduction for Severe Asthma Patients Using Health Insurance Claim Database
Acronym: HAYATE
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D3250R00092
Record Dates: First submitted 2021-10-25; First posted 2021-11-29 (Actual); Last update posted 2023-03-17 (Actual); Status verified 2023-03

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

SUMMARY:
This study is a retrospective cohort study of patients diagnosed with asthma based on the data extracted from the MDV database. The study period is from 1st Jun 2016 to 29th February 2020 .

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged ≥16 years at index date.
2. Patients with records of receiving high dose ICS or high dose ICS/LABA and diagnosed as asthma (ICD-10 code: J45 or J46 ) during baseline period. High dose ICS and high dose ICS/LABA will be defined in the appendices (Table 6-9).
3. Patients who had visit histories at least one visit during baseline period, at least two visits during outcome period and at least one visit after outcome period.
4. Patients who had a total of 12 weeks of OCS prescribed during the baseline period including the index date.

Exclusion Criteria:

1. Patients diagnosed with selected autoimmune diseases during the baseline period because OCS is used as a therapeutic agent for these disease. Autoimmune disease will be identified by following ICD-10 code (M30, M05, M06, L93, M32, K50, K51, K52, N04).

Ages: 16 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All individuals who meet followed inclusion / exclusion criteria will be identified between study period in the MDV database, and will be included in Full Analysis Set.
Sampling Method: Probability Sample
Enrollment: 2927 (Actual)
Dates: Start 2022-01-06 (Actual); Primary Completion 2022-05-16 (Actual); Study Completion 2022-05-16 (Actual)

PRIMARY OUTCOMES:
Percentage reduction on daily dose of maintenance OCS from week-0 to week-24 | from week-0 to week-24
Percentage of patients who achieved >0%, ≥25%, ≥50%, 100% OCS reduction of daily maintenance OCS dose from week-0 to week-24 respectively. | from week-0 to week-24
  (the number of patients who achieved >0%, ≥25%, ≥50%, 100% OCS reduction of daily maintenance OCS dose) / (number of total patients ) x 100
Total amount of maintenance OCS prescribed during outcome period. | from index date to 24 weeks later
Percentage reduction on daily dose of maintenance OCS from week-0 to week-24 with two groups. | from week-0 to week-24
  Two groups are amount of regular OCS use at index date is ①5mg/day or more and ②10mg/day or more respectively.
Total amount of SCS during outcome period. | from index date to 24 weeks later

SECONDARY OUTCOMES:
Percentage of OCS reduction of maintenance OCS dose from week-0 to week-8. | from week-0 to week-8.
Percentage of OCS reduction of maintenance OCS dose from week-0 to week-16. | from week-0 to week-16

OTHER OUTCOMES:
Percentage reduction on daily dose of maintenance OCS from week-0 to week-24 between benralizumab or mepolizumab initiated severe asthma patients with regular maintenance OCS use and BIO non-initiated severe asthma patients with regular. | from week-0 to week-24
Total amount of maintenance OCS prescribed during one year and two years respectively. | during one year and two years
Total amount of SCS during one year and two year respectively. | during one year and two years
Percentage of patients with an exacerbation during outcome period. | from index date to 24 weeks later
Percentage of patients with no exacerbation during outcome period. | from index date to 24 weeks later
Annualized exacerbation rate. | from index date to 24 weeks later
Percentage of patients who used asthma related medication during baseline period and outcome period respectively. | during baseline period and outcome period
The total canisters of SABA prescribed during baseline period and outcome period respectively. | during baseline period and outcome period
Percentage of patients who received high dose ICS or high dose ICS/LABA during outcome period. | from index date to 24 week later

CONTACTS AND LOCATIONS:
Locations (1):
- Research Site, Tokyo, Japan

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials/studies via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract fordata accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- [Derived] Tanaka A, Takahashi M, Fukui A, Arita Y, Fujiwara M, Makita N, Tashiro N. Oral Corticosteroid Reduction Between Biologics Initiated and Non-Initiated Patients with Severe Asthma. J Asthma Allergy. 2023 Aug 14;16:839-849. doi: 10.2147/JAA.S411404. eCollection 2023. PMID 37600852
- See also: Related Info — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D3250R00092&attachmentIdentifier=11d3b05b-eaaa-44ef-90fb-e668e980e61d&fileName=HAYATE_Study_report_synopsis.pdf&versionIdentifier=